CLINICAL TRIAL: NCT00082472
Title: Phase I/II Study of Inhaled Doxorubicin Plus IV Docetaxel and Cisplatin in Patients With Locally Advanced or Metastatic Unresectable Non Small Cell Lung Cancer
Brief Title: Inhaled Doxorubicin Plus IV Docetaxel and Cisplatin in Patients With Non-Small-Cell Lung Carcinoma (NSCLC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zivena (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dox-2a-07
Record Dates: First submitted 2004-05-11; First posted 2004-05-12 (Estimated); Last update posted 2006-04-18 (Estimated); Status verified 2006-04

CONDITIONS: NSCLC
Keywords: NSCLC; Metastatic; Unresectable; No Prior Chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Docetaxel; Cisplatin

INTERVENTIONS:
Drug: Doxorubicin HCl Inhalation Solution
Drug: Docetaxel
Drug: Cisplatin

SUMMARY:
This study is intended to show whether inhaled chemotherapy can be added to a standard IV chemotherapy regime, to investigate the additional toxicities and to show initial evidence of efficacy of the combination.

DETAILED DESCRIPTION:
Primary Objective of Phase I

* To determine the maximal and Phase II dose of inhaled doxorubicin HCl when given in combination with IV docetaxel and cisplatin in patients with locally advanced or metastatic unresectable NSCLC who have not been previously treated with chemotherapy.

Primary Objective of Phase II

* To obtain preliminary evidence of therapeutic activity using imaging studies in patients with measurable or evaluable lung lesions and serial measurements of disease-related pulmonary symptoms and pulmonary function.

Secondary Objective

* To define the nature of the toxic effects of inhaled doxorubicin when given in combination with IV docetaxel and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic proof of locally advanced or metastatic unresectable NSCLC, Patients with the pneumonic form of BAC, or cavitary lesions > 3.5 cm or with cavitary lesions of any size with air/fluid levels are not eligible.
* No prior chemotherapy or biologic therapy for lung cancer
* Measurable or evaluable pulmonary disease required
* Age > 18 years
* ECOG performance status of 0-1
* Adequate bone marrow, hepatic, and renal function
* Total bilirubin < ULN
* SGOT and/or SGPT may be up to 2.5 x ULN if alkaline phosphatase is ≤ ULN, or alkaline phosphatase may be up to 4 x ULN if SGOT and SGPT are both ≤ ULN
* Creatinine <1.5 mg/dL or creatinine clearance > 60 mL/min/1.7 m2 BSA
* Patients must have the following pulmonary function test values:

  * DLCO > 50% predicted. (DLCO must be adjusted for the patient's hemoglobin)
  * FVC> 50% of predicted
  * FEV1 >50% of predicted
  * Resting oxygen saturation > 90%
  * Exercise oxygen saturation > 85%
* Prior surgery is permitted provided full recovery has occurred
* Patients may not have received prior radiotherapy to the lungs. Patients with only chest wall or breast irradiation are eligible provided there is no radiographic evidence of pulmonary damage attributed to radiation therapy. Patients who have undergone Radioactive Iodine (RAI) therapy are also eligible.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.

Exclusion Criteria:

* Women must not be pregnant or breast-feeding during this study. Men and women with reproductive potential must use an effective contraceptive method while on this study and agree to use an effective method for three months after completing chemotherapy.
* Patients with large obstructive pulmonary lesions that may cause blockage of delivery of aerosolized drug to the affected lung, in the judgment of the treating physician. A ventilation scan is recommended if the status is unclear.
* Patients with other active malignancies. Patients with a history of prior malignancy other than NSCLC must not have received chemotherapy within the past 5 years and may not have had prior therapy with mitomycin (> 25 mg/m2), bleomycin or nitrosoureas (> 200 mg/m2). The patient may not have had any indication of pulmonary toxicity from the chemotherapy.
* Serious active infections which are not controlled such that the patient continues to manifest symptoms despite treatment
* Patients with progressive extra-pulmonary metastases who are unlikely to benefit from systemic or inhaled chemotherapy, e.g., extensive liver metastases, untreated brain metastases or treated brain metastases which are not clinically stable. If patients have received radiation treatment for brain metastases, at least 3 weeks must have elapsed since the last treatment and the patient must have recovered from all toxicity, not be receiving corticosteroids and have stable neurologic function off corticosteroids.
* Patients with known hypersensitivity to platinum compounds or taxanes or other drugs formulated with polysorbate 80
* asthma
* uncontrolled diabetes mellitus
* Patients who have undergone lung transplantation
* unstable angina, congestive heart failure, or symptomatic arrhythmias or any other serious illness or medical condition that in the judgment of the investigator compromises the patient's safety
* clinically significant neuropathy (≥ Grade 1) by history or physical examination
* Patients using other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-01

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Yale University Cancer Center, New Haven, Connecticut
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - Arthur G James Cancer Hospital and Richard Solove Research Institute at Ohio State University, Columbus, Ohio
  - University of Wisconsin Cancer Center, Madison, Wisconsin